CLINICAL TRIAL: NCT02470338
Title: A Single-Blinded Randomized Controlled Trial Comparing Modified Brostrӧm Procedure With and Without Diagnostic Arthroscopy for Treatment of Lateral Ankle Instability
Brief Title: Modified Brostrӧm Procedure With and Without Possible Arthroscopy for Lateral Ankle Instability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn as researcher left
Sponsor: Edna Rath (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Edna Rath, Human Protection Director, William Beaumont Army Medical Center
Organization: William Beaumont Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 404631-1
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lateral Ankle Instability
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBP plus ankle arthroscopy (Group A) (Active Comparator): Group A will receive a diagnostic ankle arthroscopy followed by the Modified Brostrӧm Procedure (MBP). In the ankle arthroscopy, multiple pictures are taken inside of the joint to note possible pathologic processes (for example - osteochondral lesions of the talus). Ankle arthroscopy involves one incision in the middle of the ankle anteriomedial (middle) incision and one incision on the outside of the ankle. Each incision (a small cut in the skin) is roughly 5mm in length (which is about 0.2 inches). After the incision is made, the participant will receive a diagnostic ankle arthroscopy.If the surgeon detects an abnormality inside the joint, he will operate on the abnormality with the arthroscope according to the generally accepted principles for treating the abnormality.
  Interventions: Procedure: MBP plus arthroscopy (Group A)
- MBP alone (Group B) (Sham Comparator): Group B will receive sham skin incisions on the ankle a Modified Brostrӧm Procedure (MBP) alone (that is, there will be no diagnostic ankle arthroscopy) followed by the Modified Brostrӧm Procedure (MBP). If a participant is assigned to Group B, the participant will receive two small superficial skin incisions at the sites where the investigators would normally insert instruments for the ankle arthroscopy. As with Group A, there will be one anteriomedial (middle) incision on the middle of the ankle and one anteriolateral (side) incision to on the outside of the ankle. Each incision will be roughly 5mm in length and 5 mm in depth, but will not violate subcutaneous tissue. The width of these incisions will be the width of the blade, at 1mm. However, unlike Group A, the participants in Group B will not have any instruments inserted into their ankle and will not have any operation to repair or remove damaged tissue.
  Interventions: Procedure: MBP alone (Group B)

INTERVENTIONS:
Procedure: MBP plus arthroscopy (Group A)
  Arms: MBP plus ankle arthroscopy (Group A)
Procedure: MBP alone (Group B)
  Arms: MBP alone (Group B)

SUMMARY:
This study is to show that the investigators believe the Modified Brostrӧm Procedure (MBP) can be completed without a routine ankle arthroscopy. Routine ankle arthroscopy, if determined not to be necessary in all cases, is a waste of resources in terms of operating room, surgeon, and staff time as well causing an increase in hospital financial expenses. Most importantly, this procedure is morbid. Ankle arthroscopy forces a patient's foot into distraction for up to one hour, exposes the patient to potentially longer anesthesia exposure that is unnecessary, increases infectious risks, and requires exposure at the portal sites near superficial nerves.

DETAILED DESCRIPTION:
The purpose of this investigation is to determine if ankle arthroscopy is necessary in the treatment of routine ankle instability without evidence of intra-articular pathology on MRI. Our study population will include those individuals whose ankle MRI is inconclusive or negative for intra-articular pathologies, and intra-articular ankle pain is not a predominant presenting symptom. Although it is our current practice at WBAMC not to conduct an ankle arthroscopy on this group of patients, there is a debate in the literature on whether the arthroscopy should be conducted. Thus, the purpose of this study is to examine the MBP with and without ankle arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to independently consent for surgery
2. Able to demonstrate an understanding of study procedures
3. Adult patient 18 years of age or older
4. All active duty soldiers, Veterans, dependents
5. Ability to comply with study procedures for the entire length of the study
6. Presence of lateral ankle instability meeting operative criteria listed in 6.2.1 with documented failed conservative measures such as: physical therapy, ankle braces, and rest

Exclusion Criteria:

1. Unable to obtain medical clearance for surgery
2. Recent (1 month) febrile illness that precludes or delays participation
3. History of or suspected of drug/alcohol abuse, as these patients may not be compliant with physical therapy. All patients are required to be immobilized for 6 weeks after surgery
4. Pregnant women, this is an elective procedure and a MBP or ankle arthroscopy is not typically offered to pregnant women. Screening for pregnancy is done as part of standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Talar Tilt Exam | Changes in Talar Tilt Exam scores from initial pre-op through the end of study. (Pre- Operative, Day of Surgery, Post-Op Month 3, Post Op Month 6, Post Op Month 12, Post Op Month 24)
  the angle formed by the tibial plafond and talar dome is measured as inversion force is applied to the hindfoot at 10-20 degrees of plantarflexion. A tilt of 0-23 degrees is considered normal though most ankles measure 0-5 degrees.
Anterior Drawer Exam | Changes in Anterior Drawer Exam scores from initial pre-op through the end of study. (Pre- Operative, Day of Surgery, Post-Op Month 3, Post Op Month 6, Post Op Month 12, Post Op Month 24)
  a test in which a patient is seated with the knee flexed, and the tibia is fixed with one hand while the ankle is grasped with the other hand, plantarflexed 10 degrees, and the talus is translated anteriorly under fluoroscopy. The degree of translation in mm is measured. To put this in perspective, a translation of >8mm is considered diagnostic for an anterior talofibular ligament (ATFL) tear.
Visual Analog Scale | Changes in Visual Analog Scale scores from initial pre-op through the end of study. (Pre- Operative, Day of Surgery, Post-Op Month 3, Post Op Month 6, Post Op Month 12, Post Op Month 24)
  a psychometric response scale in which a patient indicates their agreement with a statement along a continuous line. In our case, we will record how satisfied the patient is with their outcome/present post-operative state on a scale of 1-100.
American Orthopaedic Foot and Ankle Society | Changes in American Orthopaedic Foot and Ankle Society scores from initial pre-op through the end of study. (Pre- Operative, Day of Surgery, Post-Op Month 3, Post Op Month 6, Post Op Month 12, Post Op Month 24)
  Hindfoot Score is a subjective outcome scale evaluating pain, function, and alignment

CONTACTS AND LOCATIONS:
Overall Officials: MAJ Justin D Orr, MD, MC, USA, Principal Investigator — Program Director
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buchbinder R, Osborne RH, Ebeling PR, Wark JD, Mitchell P, Wriedt C, Graves S, Staples MP, Murphy B. A randomized trial of vertebroplasty for painful osteoporotic vertebral fractures. N Engl J Med. 2009 Aug 6;361(6):557-68. doi: 10.1056/NEJMoa0900429. PMID 19657121
- [Background] DiGiovanni CW, Brodsky A. Current concepts: lateral ankle instability. Foot Ankle Int. 2006 Oct;27(10):854-66. doi: 10.1177/107110070602701019. No abstract available. PMID 17054892
- [Background] DIGiovanni BF, Fraga CJ, Cohen BE, Shereff MJ. Associated injuries found in chronic lateral ankle instability. Foot Ankle Int. 2000 Oct;21(10):809-15. doi: 10.1177/107110070002101003. PMID 11128010
- [Background] 4. Kitaoka HB. The Foot and Ankle. Master Techniques in Orthopaedic Surgery. 2013. 3rd edition: 515-536. Lippincott Williams & Wilkins. Philadelphia, PA.
- [Background] Komenda GA, Ferkel RD. Arthroscopic findings associated with the unstable ankle. Foot Ankle Int. 1999 Nov;20(11):708-13. doi: 10.1177/107110079902001106. PMID 10582846
- [Background] Maffulli N, Ferran NA. Management of acute and chronic ankle instability. J Am Acad Orthop Surg. 2008 Oct;16(10):608-15. doi: 10.5435/00124635-200810000-00006. PMID 18832604
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735
- [Background] O'Neill PJ, Van Aman SE, Guyton GP. Is MRI adequate to detect lesions in patients with ankle instability? Clin Orthop Relat Res. 2010 Apr;468(4):1115-9. doi: 10.1007/s11999-009-1131-0. Epub 2009 Oct 23. PMID 19851818
- [Background] Richardson EG. Orthopaedic Knowledge Update 3. 2004. American Academy of Orthopaedic Surgeons. Rosemont, IL.
- [Background] Sihvonen R, Paavola M, Malmivaara A, Itala A, Joukainen A, Nurmi H, Kalske J, Jarvinen TL; Finnish Degenerative Meniscal Lesion Study (FIDELITY) Group. Arthroscopic partial meniscectomy versus sham surgery for a degenerative meniscal tear. N Engl J Med. 2013 Dec 26;369(26):2515-24. doi: 10.1056/NEJMoa1305189. PMID 24369076
- [Background] van Dijk CN, Bossuyt PM, Marti RK. Medial ankle pain after lateral ligament rupture. J Bone Joint Surg Br. 1996 Jul;78(4):562-7. PMID 8682821